CLINICAL TRIAL: NCT05516862
Title: Determining the Right Acupuncture for Good Recovery Over Neuropsychiatric Trauma (DRAGON)
Brief Title: Determining the Right Acupuncture for Good Recovery Over Neuropsychiatric Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Crawford (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Paul Crawford, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USUHS.2022-101
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: PTSD; Post Traumatic Stress Disorder; Acupuncture
Keywords: PTSD; DRAGONS; family medicine residency
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Script followed by Dragons Acupuncture (external Dragons points with patient prone for 15 minutes followed by internal Dragons points with patient supine for 15 minutes).
  Interventions: Other: Dragons acupuncture
- Group 2 (Sham Comparator): Script followed by Dragons sham acupressure placed at the Dragons points (external Dragons points with patient prone for 15 minutes followed by internal Dragons points with patient supine for 15 minutes).
  Interventions: Other: Dragons acupressure
- Group 3 (Placebo Comparator): Script followed by Acupuncturist lightly touching Dragons points (external Dragons points with patient prone for 15 minutes followed by internal Dragons points with patient supine for 15 minutes).
  Interventions: Other: Dragons placebo

INTERVENTIONS:
Other: Dragons acupuncture — The treatment we are studying is supposed to help the rational and emotional brain effectively communicate, so that the emotional brain can finally realize the trauma experienced is no longer a threat. We call this re-processing. It does not take away the memory but it allows the rational brain to see the memory as just a memory without the emotional brain initiating your fight, flight or freeze system. This allows the mind to take the file off the messy desk and put it away. The treatment was named by the Chinese and is called "External and Internal Dragons". According to the Chinese, the External Dragons represent all the bad (traumatic) things that happen to us. The Internal Dragons live inside us, and fight off the External Dragons.
  Subject will lay on your stomach and have 7 needles placed in head, upper back, lower back and ankles.
  Arms: Group 1
Other: Dragons acupressure — The treatment we are studying is supposed to help the rational and emotional brain effectively communicate, so that the emotional brain can finally realize the trauma experienced is no longer a threat. We call this re-processing. It does not take away the memory but it allows the rational brain to see the memory as just a memory without the emotional brain initiating your fight, flight or freeze system. This allows the mind to take the file off the messy desk and put it away. The treatment was named by the Chinese and is called "External and Internal Dragons". According to the Chinese, the External Dragons represent all the bad (traumatic) things that happen to us. The Internal Dragons live inside us, and fight off the External Dragons.
  Subject will lay on your stomach and have 7 small acupressure adhesive bandages placed on head, upper back, lower back and ankles.
  Arms: Group 2
Other: Dragons placebo — The treatment we are studying is supposed to help the rational and emotional brain effectively communicate, so that the emotional brain can finally realize the trauma experienced is no longer a threat. We call this re-processing. It does not take away the memory but it allows the rational brain to see the memory as just a memory without the emotional brain initiating your fight, flight or freeze system. This allows the mind to take the file off the messy desk and put it away. The treatment was named by the Chinese and is called "External and Internal Dragons". According to the Chinese, the External Dragons represent all the bad (traumatic) things that happen to us. The Internal Dragons live inside us, and fight off the External Dragons.
  Subject will lay on your stomach and the doctor will touch 7 points on head, upper back, lower back and ankles.
  Arms: Group 3

SUMMARY:
This study seeks to verify that a specific acupuncture treatment is effective at reducing symptoms of neuropsychiatric trauma found in those diagnosed with Post-Traumatic Stress Disorder (PTSD).

DETAILED DESCRIPTION:
Traumatic stress experienced by service members negatively affects their ability to psychologically and emotionally cope with operational and family stressors. Physically, chronic pain complaints are higher in those with neuropsychiatric trauma. These can lead to a decrease in quality and duration of life. The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) classifies Post-Traumatic Stress Disorder as an anxiety disorder (DSM). To achieve this diagnosis a person must be exposed to a traumatic event and then experience long lasting intrusive symptoms such as nightmares, irritability, flashbacks and trauma related thoughts or feelings that impair their ability to function in their day-to-day activities. These symptoms can be very distressing to individuals, often leading to other mental health disorders such as depression and generalized anxiety. They also frequently have widespread negative effects on their families, friends, co-workers and ultimately the mission of the United States Military. A leading theory regarding the underlying cause of PTSD states that the sympathetic nervous system (fight or flight) is upregulated every time the emotional centers of the brain are reminded of the traumatic event. This upregulation causes symptoms listed above along with physiologic symptoms such as elevations in heart rate, breathing and blood pressure. This can occur even in the absence of the conscious mind recognizing what is triggering this sympathetic response1.

The overall effect for a patient is the overwhelming feeling that a terrifying traumatic event experienced many years ago is happening again in the present. Treatments aimed at downregulation of the sympathetic nervous system are common; however, treatments that can "break" the connection between prior trauma, the emotional centers of the brain and the sympathetic nervous system have the potential to treat the true underlying cause of PTSD.

Treatment of psychological, emotional, and physical symptoms of Post-Traumatic Stress Disorder (PTSD) can include medication, psychotherapy, or some combination of the two. Evidence supports the idea that receiving traditional treatment for PTSD symptoms such as psychotherapy is something that many veterans are disinclined to do due to a perceived stigma of admitting that they have a mental illness (Mittal); although when adhered to, psychotherapy can cause significant improvement in PTSD symptoms such as sleep disturbance, depression, and suicidality 2. Alternatives to these traditional therapies are needed.

Compared to traditional CBT, acupuncture offers a treatment effect for PTSD similar to CBT (Hollifield)6. A systematic review and meta-analysis examining prospective controlled clinical trials found no statistical difference between acupuncture and CBT (Kim)7. Compared to traditional SSRIs, acupuncture may be a treatment option for those experiencing SSRI side effects of sexual dysfunction, weight gain, and sleep disturbance (Kim)7. One part of Acupuncturists Without Borders (AWB) reports that veterans given acupuncture for PTSD reported better sleep with fewer nightmares, a clearer mental state, and less stress (Sneizck)8. Auricular (ear) acupuncture treatments in the veteran and servicemember population diagnosed with PTSD found that those treated had improved sleep, increased relaxation, decreased pain, and improvements in depression symptoms (Huang; Engel; King)9,10,11.

Veterans also reacted favorably to the concept of the brief course of auricular acupuncture treatments, especially those who had avoided PTSD treatment due to associated stigma or lack of faith in traditional methods (King)11.

There is an urgent need for additional, empirically validated, non-opioid alternative strategies attached to less stigma for symptoms associated with PTSD. Programs across the United States military are showing the effect of integrative medicine approaches, and this study will serve as another building block in the emerging whole person approach to military medicine12.

One path to successful PTSD treatments may involve the vagal nerve. The vagal nerve is responsible for connecting the brain's central functions with peripheral organ function all throughout the body and counteracts the sympathetic response ( creating a rest and digest response)13. It regulates the body's stress response; dysregulation of the vagus-controlled hypothalamic-pituitary-adrenal axis is connected to PTSD14. Accordingly, external stimulus to the vagal nerve could forcefully alleviate dysregulation15. Historically, vagal nerve stimulation was achieved through surgical device implantation. Noninvasive vagal nerve stimulation methods are being newly developed and can positively affect a variety of physiologic processes (Bremner)13.

We suggest that our acupuncture protocol is another novel method that can stimulate parts of the vagal nerve.

MicroRNA biomarkers for posttraumatic stress disorder: MicroRNAs (miRNAs, miRs) are small RNA molecules (~ 22 nucleotides long) and are often, but need not be, post-transcriptional regulators that bind to complementary sequences on target messenger RNA transcripts (mRNA), usually resulting in translational repression and gene silencing. MiRNA may serve as good biomarkers because they are highly stable in serum due to their ability to withstand repeated freeze thaw, enzymatic degradation, and extreme pH conditions.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty members and DoD beneficiaries(i.e. former military, spouse, dependent child), 18-65 years old
* Meeting the criteria for PTSD based on PCL-5 (past month scores) score of 31 or higher
* At least 1 positive response to at least one item on the LEC-5.

Exclusion Criteria:

* Pregnant, may be pregnant, or attempting to become pregnant. There areno known risks of this acupuncture in pregnant patients; however, we will exclude pregnancy due to the location of the needles (right over the uterus in 3rd trimester) and risk of exacerbating anxiety that may cause stress on the baby. Subjects will be told to let us know if they become pregnant so we can disenroll them from the study.
* Prior treatment with Dragons acupuncture
* History of hospitalization for mental health reasons within the last year
* Active Suicidal thoughts (is currently considering suicide or has a plan) or suicide attempt within the last year. This will be assessed by direct questioning.
* Is currently receiving acupuncture or other non-medication treatments specifically for PTSD (patients can elect to forgo PTSD treatments during the study period and then resume after the study period is over; ie halt therapy during the study period)
* Legally Authorized Representatives will not be utilized in this study

**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | visit 1 (week 0)
  The CAPS-5 is a structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week. The CAPS-5 will be applied for its first purpose in this study. The instrument produces a total symptom severity score by summing severity scores for the 20 DSM-5 PTSD symptoms and symptom cluster severity scores calculated by summing individual item severity scores for symptoms corresponding to a given DSM-5 cluster. There are five symptom cluster severity scores: Criterion B, Criterion C, Criterion D, Criterion E and Criterion disassociation.
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | visit 6 (week 8)
  The CAPS-5 is a structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week. The CAPS-5 will be applied for its first purpose in this study. The instrument produces a total symptom severity score by summing severity scores for the 20 DSM-5 PTSD symptoms and symptom cluster severity scores calculated by summing individual item severity scores for symptoms corresponding to a given DSM-5 cluster. There are five symptom cluster severity scores: Criterion B, Criterion C, Criterion D, Criterion E and Criterion disassociation.
PTSD checklist for DSM-5 (PCL-5) | visit 1 (week 0)
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.
PTSD checklist for DSM-5 (PCL-5) | visit 3 (week 2)
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.
PTSD checklist for DSM-5 (PCL-5) | visit 4 (week 3)
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.
PTSD checklist for DSM-5 (PCL-5) | visit 5 (week 4)
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.
PTSD checklist for DSM-5 (PCL-5) | visit 6 (week 8)
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.

SECONDARY OUTCOMES:
microRNA biomarkers | visit 1 (week 0)
  Changes in microRNA (miRNA) serum biomarkers miRNA-518f-3p, miRNA-486-5p, miRNA-let-7b, miRNA-220, and miRNA-433.
microRNA biomarkers | visit 6 (week 8)
  Changes in microRNA (miRNA) serum biomarkers miRNA-518f-3p, miRNA-486-5p, miRNA-let-7b, miRNA-220, and miRNA-433.

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data.

REFERENCES:
- [Background] Van, K. B. A. (2014). The body keeps the score: Brain, mind, and body in the healing of trauma. p 44-46
- [Background] Vitale A, Byma L, Sun S, Podolak E, Wang Z, Alter S, Galfalvy H, Geraci J, Langhoff E, Klingbeil H, Yehuda R, Haghighi F, Feder A. Effectiveness of Complementary and Integrative Approaches in Promoting Engagement and Overall Wellness Toward Suicide Prevention in Veterans. J Altern Complement Med. 2021 Mar;27(S1):S14-S27. doi: 10.1089/acm.2020.0245. PMID 33788604
- [Background] Jiang Y, Hao Y, Zhang Y, Liu J, Wang X, Han J, Fang J, Zhang J, Cui C. Thirty minute transcutaneous electric acupoint stimulation modulates resting state brain activities: a perfusion and BOLD fMRI study. Brain Res. 2012 May 31;1457:13-25. doi: 10.1016/j.brainres.2012.03.063. Epub 2012 Apr 3. PMID 22541167
- [Background] Xiang XH, Chen YM, Zhang JM, Tian JH, Han JS, Cui CL. Low- and high-frequency transcutaneous electrical acupoint stimulation induces different effects on cerebral mu-opioid receptor availability in rhesus monkeys. J Neurosci Res. 2014 May;92(5):555-63. doi: 10.1002/jnr.23351. Epub 2014 Jan 31. PMID 24482187
- [Background] Feng B, Zhang Y, Luo LY, Wu JY, Yang SJ, Zhang N, Tan QR, Wang HN, Ge N, Ning F, Zheng ZL, Zhu RM, Qian MC, Chen ZY, Zhang ZJ. Transcutaneous electrical acupoint stimulation for post-traumatic stress disorder: Assessor-blinded, randomized controlled study. Psychiatry Clin Neurosci. 2019 Apr;73(4):179-186. doi: 10.1111/pcn.12810. Epub 2019 Jan 22. PMID 30565342
- [Background] Hollifield M. Acupuncture for posttraumatic stress disorder: conceptual, clinical, and biological data support further research. CNS Neurosci Ther. 2011 Dec;17(6):769-79. doi: 10.1111/j.1755-5949.2011.00241.x. Epub 2011 Feb 26. PMID 22070661
- [Background] Kim YD, Heo I, Shin BC, Crawford C, Kang HW, Lim JH. Acupuncture for posttraumatic stress disorder: a systematic review of randomized controlled trials and prospective clinical trials. Evid Based Complement Alternat Med. 2013;2013:615857. doi: 10.1155/2013/615857. Epub 2013 Feb 6. PMID 23476697
- [Background] Sniezek DP. Community-Based Wounded Warrior Sustainability Initiative (CBWSI): an integrative medicine strategy for mitigating the effects of PTSD. J Rehabil Res Dev. 2012;49(3):ix-xix. doi: 10.1682/jrrd.2012.02.0025. No abstract available. PMID 22773206
- [Background] Huang W, Johnson TM, Kutner NG, Halpin SN, Weiss P, Griffiths PC, Bliwise DL. Acupuncture for Treatment of Persistent Disturbed Sleep: A Randomized Clinical Trial in Veterans With Mild Traumatic Brain Injury and Posttraumatic Stress Disorder. J Clin Psychiatry. 2018 Dec 11;80(1):18m12235. doi: 10.4088/JCP.18m12235. PMID 30549498
- [Background] Engel CC, Cordova EH, Benedek DM, Liu X, Gore KL, Goertz C, Freed MC, Crawford C, Jonas WB, Ursano RJ. Randomized effectiveness trial of a brief course of acupuncture for posttraumatic stress disorder. Med Care. 2014 Dec;52(12 Suppl 5):S57-64. doi: 10.1097/MLR.0000000000000237. PMID 25397825
- [Background] King CH, Moore LC, Spence CD. Exploring Self-Reported Benefits of Auricular Acupuncture Among Veterans With Posttraumatic Stress Disorder. J Holist Nurs. 2016 Sep;34(3):291-9. doi: 10.1177/0898010115610050. Epub 2015 Nov 3. PMID 26530240
- [Background] Hull A, Brooks Holliday S, Eickhoff C, Sullivan P, Courtney R, Sossin K, Adams A, Reinhard M. Veteran participation in the integrative health and wellness program: Impact on self-reported mental and physical health outcomes. Psychol Serv. 2019 Aug;16(3):475-483. doi: 10.1037/ser0000192. Epub 2018 Apr 5. PMID 29620393
- [Background] Bremner JD, Gurel NZ, Wittbrodt MT, Shandhi MH, Rapaport MH, Nye JA, Pearce BD, Vaccarino V, Shah AJ, Park J, Bikson M, Inan OT. Application of Noninvasive Vagal Nerve Stimulation to Stress-Related Psychiatric Disorders. J Pers Med. 2020 Sep 9;10(3):119. doi: 10.3390/jpm10030119. PMID 32916852
- [Background] de Kloet CS, Vermetten E, Geuze E, Kavelaars A, Heijnen CJ, Westenberg HG. Assessment of HPA-axis function in posttraumatic stress disorder: pharmacological and non-pharmacological challenge tests, a review. J Psychiatr Res. 2006 Sep;40(6):550-67. doi: 10.1016/j.jpsychires.2005.08.002. Epub 2005 Oct 7. PMID 16214171
- [Background] Thrivikraman KV, Zejnelovic F, Bonsall RW, Owens MJ. Neuroendocrine homeostasis after vagus nerve stimulation in rats. Psychoneuroendocrinology. 2013 Jul;38(7):1067-77. doi: 10.1016/j.psyneuen.2012.10.015. Epub 2012 Nov 16. PMID 23159723